CLINICAL TRIAL: NCT03048539
Title: Comparison of Quality of Life Between Patients Underwent Transoral Endoscopic Thyroid Surgery and Conventional Surgery
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Khon Kaen University (Other)
Responsible Party: Principal Investigator, Pornthep Kasemsiri, Principal investigator, Khon Kaen University
Other Study IDs: HE591505
Record Dates: First submitted 2017-02-02; First posted 2017-02-09 (Estimated); Last update posted 2017-03-07 (Actual); Status verified 2017-03

CONDITIONS: Quality of Life; Transoral Endoscopic Thyroidectomy; Conventional Thyroidectomy
Keywords: Endoscopic surgery; Thyroidectomy; Quality of life

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Transoral endoscopic thyroidectomy: Patient who fit with the eligible criteria and choose endoscopic thyroidectomy by himself.
  Interventions: Procedure: Transoral endoscopic thyroidectomy
- Conventional thyroidectomy: Patient who fit with the eligible criteria and choose conventional thyroidectomy by himself.

INTERVENTIONS:
Procedure: Transoral endoscopic thyroidectomy — This procedure will remove thyroid lobe through oral vestibule. Aim to avoid scar at anterior neck.
  Groups: Transoral endoscopic thyroidectomy

SUMMARY:
The purpose of this study is to determine the quality of life of transoral endoscopic thyroidectomy compare with open thyroidectomy, Furthermore, postoperative complication will be assessed, also.

DETAILED DESCRIPTION:
Regarding type of surgery, doctor will just advice about risk and benefit of any type of surgery. And then patient will select by himself. Patients are not assigned to endoscopic or conventional group.

This study start to enrolled patients after surgery. And the quality of life will be observed at 2, 6 and 12 weeks, respectively.

ELIGIBILITY:
Inclusion Criteria:

* Patient who underwent thyroid lobectomy for benign thyroid nodule less or equal 5 cm

Exclusion Criteria:

* previous neck surgery
* suspected thyroid carcinoma
* patient who failure endoscopic thyroidectomy and change to conventional surgery

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Patient who underwent thyroid lobectomy
Sampling Method: Non-Probability Sample
Enrollment: 38 (Estimated)
Dates: Start 2017-02-06 (Actual); Primary Completion 2019-12-31 (Estimated); Study Completion 2019-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in quality of life after surgery | 2,6,12 weeks
  Quality of life will assessed by Short form health survey 36 and specific questionnaire for thyroidectomy. These questionnaires will assess at 2,6 and 12 weeks after surgery. The quality of life results (6 and 12 weeks) will be observed that change from 2 weeks after surgery. Furthermore, investigators will compare score of Short form health survey 36 and specific quality of life questionnaire for thyroidectomy between endoscopic and open technique at 2,6,12 week after surgery, also.

SECONDARY OUTCOMES:
Postoperative complication | 2,6, and 12 weeks
  The complications will assess at 2,6, and 12 week after surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Pornthep Kasemsiri, MD, Principal Investigator — Khon Kaen University
Locations (1):
- Khon Kaen University, Khon Kaen, Changwat Khon Kaen, Thailand

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Anuwong A. Transoral Endoscopic Thyroidectomy Vestibular Approach: A Series of the First 60 Human Cases. World J Surg. 2016 Mar;40(3):491-7. doi: 10.1007/s00268-015-3320-1. PMID 26546193
- [Derived] Kasemsiri P, Trakulkajornsak S, Bamroong P, Mahawerawat K, Piromchai P, Ratanaanekchai T. Comparison of quality of life between patients undergoing trans-oral endoscopic thyroid surgery and conventional open surgery. BMC Surg. 2020 Jan 29;20(1):18. doi: 10.1186/s12893-020-0685-3. PMID 31996201